CLINICAL TRIAL: NCT01543919
Title: A Phase 2B, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Once-Daily Orally Administered PH-797804 For 12 Weeks In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD) On A Background Of Tiotropium Bromide
Brief Title: Study To Evaluate The Efficacy And Safety Of PH-797804 For 12 Weeks In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD) On A Background Of Tiotropium Bromide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6631033
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- PH-787904 (arm1) (Experimental)
  Interventions: Drug: PH-797804
- PH-787904 (arm2) (Experimental)
  Interventions: Drug: PH-797804
- PH-787904 (arm3) (Experimental)
  Interventions: Drug: PH-797804
- PH-787904 (arm4) (Experimental)
  Interventions: Drug: PH-797804
- PH-787904 (arm5) (Experimental)
  Interventions: Drug: PH-797804
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH-797804 — 0.25 mg oral tablet plus tiotropium bromide 18 microgram once daily for 12 weeks
  Arms: PH-787904 (arm1)
Drug: PH-797804 — 1 mg oral tablet plus tiotropium bromide 18 microgram once daily for 12 weeks
  Arms: PH-787904 (arm2)
Drug: PH-797804 — 3 mg oral tablet plus tiotropium bromide 18 microgram once daily for 12 weeks
  Arms: PH-787904 (arm3)
Drug: PH-797804 — 6 mg oral tablet plus tiotropium bromide 18 microgram once daily for 12 weeks
  Arms: PH-787904 (arm4)
Drug: PH-797804 — 10 mg oral tablet plus tiotropium bromide 18 microgram once daily for 12 weeks
  Arms: PH-787904 (arm5)
Drug: Placebo — Placebo oral tablet plus tiotropium bromide 18 microgram once daily for 12 weeks
  Arms: Placebo

SUMMARY:
PH-797804 is an oral anti-inflammatory drug that may reduce the inflammation that is associated with Chronic Obstructive Pulmonary Disease (COPD). PH-797804 will be dosed to patients with Chronic Obstructive Pulmonary Disease (COPD) to evaluate its potential safety and efficacy profile in Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including, the ages of 40 and 80 years.
* Subjects with a diagnosis, for at least 6 months, of moderate to severe COPD (GOLD) and who meet the criteria for Stage II-III disease: Subjects must have a post-bronchodilator FEV1/FVC ratio <0.7 and a post-bronchodilator FEV1 of 30 - 80% (inclusive) of the predicted value for age, height, race and sex using European Community for Coal and Steel ECCS standards or NHANES III standards.
* Subjects must have a smoking history of at least 10 pack-years* and meet one of the following criteria: They are current smokers, or they are ex-smokers who have abstained from smoking for at least 6 months.
* Subjects treated with tiotropium bromide (SPIRIVA HandiHaler) 18 microgram daily for at least 1 month prior to screening.
* Subjects must have had stable disease for at least 1 month prior to screening. During the screening and run-in phase subjects must be able to manage disease symptoms adequately with tiotropium bromide +/- salbutamol (albuterol) rescue medication (subjects should not use >10 actuations [100 microgram/actuations] daily for more than 2 consecutive days), without reliance on other therapies including oral or inhaled corticosteroids, other long-acting bronchodilators, nebulizer therapy, theophylline, roflumilast or regular oxygen.

Exclusion Criteria:

* A COPD exacerbation requiring treatment with oral steroids or hospitalization for the treatment of COPD within 3 months of screening.
* History of a lower respiratory tract infection or significant disease instability during the month preceding screening or during the time between screening and randomization.
* History or presence of respiratory failure, cor pulmonale or right ventricular failure.
* Subjects with home oxygen therapy (either PRN or long-term oxygen therapy).
* Any clearly documented history of adult asthma or other chronic respiratory disorders (eg, bronchiectasis, pulmonary fibrosis, pneumoconiosis).
* Known previous diagnosis of Hepatitis B or C or HIV infection (specific screening is not required).
* History of cancer (other than cutaneous basal cell) in the previous 5 years.
* Active or past history of GI hemorrhage of any etiology, peptic ulceration, erosive esophagitis, gastric outlet obstruction or inflammatory bowel disease.
* Regular use of aspirin at a dose greater than 325 mg/day.
* History within the previous 6 months of: myocardial infarction, cardiac arrhythmia (eg, atrial fibrillation, paroxysmal atrial fibrillation, atrial flutter, supraventricular tachycardia, ventricular tachycardia), left ventricular failure, unstable angina, coronary angioplasty, coronary artery bypass grafting (CABG) or cerebrovascular accident (including transient ischemic attacks).
* A family history of long QT syndrome.
* Presenting with: Any condition possibly affecting oral drug absorption (eg, gastrectomy or clinically significant diabetic gastroenteropathy).
* Any clinically significant skin lesions as described in Common Terminology Criteria for Adverse Events for Dermatology (CTCAE) Version 3.0.
* Any clinically significant active systemic or cutaneous infection including herpetic lesions.
* Congestive heart failure requiring treatment New York Heart Association (NYHA) Class III-IV.
* ECG abnormalities at screening or randomization, including those listed below: Subjects with pre-randomization evidence of QTcF prolongation (defined as >450 ms) at screening or baseline (Week 0) are not eligible for randomization. This assessment is based on a confirmed mean of the triplicate ECG recordings and is made by the investigator at the time of ECG collection.
* Predominant heart rhythm other than normal sinus rhythm eg, atrial fibrillation, atrial flutter, supraventricular tachycardia.
* Atrioventricular (AV) block greater than first degree.
* Resting heart rate >100 or <40 bpm.
* Evidence of previous myocardial infarction in the absence of clinical history consistent with these findings.
* Evidence of acute ischemia.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough (pre-treatment and pre-bronchodilator) Forced Expiratory Volume1 at Week 12. | Baseline, week 12

SECONDARY OUTCOMES:
Change from baseline in trough, pre-bronchodilator Forced Expiratory Volume1 at Weeks 2, 6, and 10 | Baseline, week 2, 6, and 10
Change from baseline in trough, pre-bronchodilator Forced Expiratory Volume6 at Weeks 2, 6, 10 and 12 | Baseline, week 2, 6, 10 and 12
Change from baseline in trough, pre-bronchodilator Forced Vital Capacity at Weeks 2, 6, 10 and 12 | Baseline, week 2, 6, 10 and 12
Change from baseline in trough, pre-bronchodilator Inspiratory Capacity at Weeks 2, 6, 10 and 12 | Baseline, week 2, 6, 10 and 12
Average change from baseline in trough, pre-bronchodilator Forced Expiratory Volume 1, Forced Expiratory Volume 6, Forced Vital Capacity and Inspiratory Capacity over 12 weeks treatment | Baseline, week 12
Change from baseline in post-study drug, pre-bronchodilator Forced Expiratory Volume1, Forced Expiratory Volume6, Forced Vital Capacity and Inspiratory Capacity at Weeks 0 and 12 | Baseline, week 0, 12
Change from baseline in post-study drug, post-bronchodilator Forced Expiratory Volume1, Forced Expiratory Volume6, Forced Vital Capacity and Inspiratory Capacity at Weeks 0 and 12 | Baseline, week 0, week 12
Change from baseline in Chronic Obstructive Pulmonary Disease symptoms (EXACT-PRO Daily Diary) over 12 weeks treatment. | Baseline, week 12
Change from baseline in Chronic Respiratory Questionnaire - Self Administered Standard (CRQ-SAS) at Weeks 2, 6, 10 and 12 | Baseline, week 2, 4, 6, 10 and 12
Patient Global Impression of Change at Week 12 | Baseline, week 12
Change from baseline (Baseline Dyspnea Index) in dyspnea (Transition Dyspnea Index) at Weeks 2, 6, 10 and 12 | Baseline, week 2, 4, 6, 10, and 12
Clinician Global Impression of Change at Week 12 | Baseline, week 12
Rescue bronchodilator use (per daily diary) over 12 weeks of therapy | Baseline, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (114):
- United States (36):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Jasper, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Montclair, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Williston, Florida
  - Pfizer Investigational Site, Duluth, Georgia
  - Pfizer Investigational Site, Fort Mitchell, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Midvale, Utah
- Pfizer Investigational Site, Buenos Aires, Argentina
- Bulgaria (6):
  - Pfizer Investigational Site, Rousse
  - Pfizer Investigational Site, Sevlievo
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
  - Pfizer Investigational Site, Troyan Municipality
  - Pfizer Investigational Site, Veliko Tarnovo
- Canada (6):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint Romuald, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Czechia (6):
  - Pfizer Investigational Site, Karlovy Vary
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Mělník
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Rokycany
  - Pfizer Investigational Site, Teplice
- Germany (9):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Gelnhausen
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, Schwerin
- Hungary (7):
  - Pfizer Investigational Site, Balassagyarmat
  - Pfizer Investigational Site, Budaörs
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Szeged
  - Pfizer Investigational Site, Szombathely
  - Pfizer Investigational Site, Törökbálint
- Japan (15):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Seto-shi, Aichi-ken
  - Pfizer Investigational Site, Toyota, Aichi-ken
  - Pfizer Investigational Site, Noda, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Yanagawa, Fukuoka
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Takamatsu, Kagawa-ken
  - Pfizer Investigational Site, Kawasaki-shi, Kanagawa
  - Pfizer Investigational Site, Zama, Kanagawa
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Saiki, Oita Prefecture
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Meguro-ku, Tokyo
  - Pfizer Investigational Site, Setagaya City, Tokyo
- Poland (2):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Slovakia (10):
  - Pfizer Investigational Site, Bardejov
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Humenné
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Liptovský Hrádok
  - Pfizer Investigational Site, Námestovo
  - Pfizer Investigational Site, Poprad
  - Pfizer Investigational Site, Spišská Nová Ves
  - Pfizer Investigational Site, Štúrovo
- South Africa (6):
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Gatesville, Western Cape
  - Pfizer Investigational Site, Parow, Western Cape
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Durban
  - Pfizer Investigational Site, Pretoria
- Spain (4):
  - Pfizer Investigational Site, Petrel, Alicante
  - Pfizer Investigational Site, Mérida, Badajoz
  - Pfizer Investigational Site, Salt, Girona
  - Pfizer Investigational Site, Pozuelo de Alarcón, Madrid
- Sweden (5):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Skene
- Pfizer Investigational Site, Taipei, Taiwan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631033&StudyName=Study%20To%20Evaluate%20The%20Efficacy%20And%20Safety%20Of%20PH-797804%20For%2012%20Weeks%20In%20Adults%20With%20Moderate%20To%20Severe%20Chronic%20Obstructive%20Pulmonary%20